CLINICAL TRIAL: NCT03529929
Title: Glucocorticoid Inflammation Paradox in Human Skeletal Muscle
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: withdrawn
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Melinda Sheffield-Moore, Professor, Texas A&M University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2017-0883
Record Dates: First submitted 2018-04-20; First posted 2018-05-18 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Aging
Keywords: glucocorticoids; aging; NFKB; Medrol; methylprednisolone
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Methylprednisolone (Experimental): Methylprednisolone glucocorticoid Medrol Dose Pack
  Medrol is supplied as white tablets, of 4mg each. The tablets come in a commercially produced blister pack with instructions for each day of the 6 day dosing on the packaging. Subjects will receive a standard 6-day, graded dosing regimen of methylprednisolone (24mg, 20mg, 16mg, 12mg, 8mg, and 4 mg on days 1 through 6 respectively).
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — 6 day dosing as dictated by Medrol 6 Day Dose Pack
  Other Names: Medrol Dose Pack; Medrol

SUMMARY:
In this project, we propose to investigate the metabolic consequences of glucocorticoid therapy, given orally as a 6 day Medrol Dose pack, on human skeletal muscle as measured by western blotting and PCR and skeletal muscle mitochondrial capacity as measured by High-Resolution Respirometry in healthy individuals. Medrol is an FDA approved drug with many clinical indications.

DETAILED DESCRIPTION:
Healthy male and female individuals ages 60 - 80 (n=10) will be studied before and after 6 days of treatment with self-administered daily oral methylprednisolone.

Subjects will report to the Texas A&M Human Clinical Research Facility (HCRF) for testing before (day 0) and after (day 6) methylprednisolone intervention. Each visit will consist of determination of lean and fat mass using DEXA and a single muscle biopsy. Blood will be collected (up to 15ml) at screening, baseline and the conclusion of the study to measure metabolites and hormones. Phone calls will be made to subjects mid-week (day 3) during the study period to ensure compliance and continued consent.

This will be an unblinded study. All participants will receive methylprednisolone treatment.

Therapeutic Interventions. Methylprednisolone (Medrol®) dose pack. Methylprednisolone is a glucocorticoid. Glucocorticoids are adrenocortical steroids, both naturally occurring and synthetic, which are readily absorbed from the gastrointestinal tract. Therapeutic methylprednisolone is approved for clinical use for a variety of disorders. Medrol®, the agent to be used in this study, is manufactured by Pfizer.

Medrol® is supplied as white tablets, of 4mg each. The tablets come in a commercially produced blister pack with instructions for each day of the 6 day dosing on the packaging. Subjects will receive a standard 6-day, graded dosing regimen of methylprednisolone (24mg, 20mg, 16mg, 12mg, 8mg, and 4 mg on days 1 through 6 respectively, Table 1 above). This methylprednisolone dosing regimen is commonly prescribed for the treatment of inflammation associated with a number of pathologies, including arthritic, respiratory, and neoplastic diseases. The Medrol® pack has clear instructions on how to administer the tablets and participants will be given additional instruction to ensure understanding for proper self-administration.

ELIGIBILITY:
Inclusion Criteria:

1. Ages: 60 - 80 years.
2. For men only: Eugonadal men, with a basal serum testosterone level for men within the normal range for the assay.
3. For women only: women must be post-menopausal.
4. Availability of transportation (i.e., subjects must be able to provide their own transportation to TAMU HCRF).
5. Ability to fast for 12 hours before each of the study visits

Exclusion Criteria:

1. Use of anticoagulant due to the risk of bleeding during the muscle biopsy procedure.
2. Current use or history of recent use of anabolic steroids or glucocorticoids (within 3 months).
3. Use of anti-bone-resorptive agents such as bisphosphonates, parathyroid hormone, or calcitonin.
4. Use of live virus vaccines in the past 30 days.
5. History of stroke.
6. History of angina that occurs with exertion or at rest or a myocardial infarction within the last 12 months.
7. Diagnosed systemic viral, bacterial, or fungal infections.
8. Any established major medical illness such as chronic obstructive pulmonary disease, or untreated sleep apnea.
9. Subjects with minor, acute inflammatory illnesses such as colds will be excluded until the acute illness has resolved.
10. Uncontrolled endocrine or metabolic disease (e.g. liver disease, renal disease, diabetes).
11. History or current diagnosis of type 1 or type 2 diabetes. High doses of glucocorticoids can increase insulin resistance and exacerbate diabetes.
12. Systolic blood pressure greater than or equal to 160mm Hg or a diastolic blood pressure greater than or equal to 100mm Hg on three consecutive measurements taken at one-week intervals. Glucocorticoids can cause fluid retention that could worsen uncontrolled hypertension. Subjects will be included if they are on two or less blood pressure medications and have a blood pressure below these criteria.
13. Subjects who engage in high intensity, elite training on a regular basis will be excluded. Additionally, subjects will be asked to refrain from any exercise during study week.
14. History of seizure disorder.
15. History of tuberculosis.
16. Current diagnosis of peptic ulcer disease, gastritis, or non-ulcer dyspepsia.
17. Current diagnosis of mental illness.
18. Current diagnosis of cognitive impairment.
19. Subjects with sleep disturbances.
20. Current self-reported immunosuppressive disorder.
21. Any other condition or event considered exclusionary by the PI and covering physician.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Oxidative Phosphorylation Capacity measured by high resolution tissue respirometry on day 0 | day 0
  Oxidative Phosphorylation will be measured in muscle tissue using high resolution respirometry (Oroboros O2K) on day 0.
Oxidative Phosphorylation Capacity measured by high resolution tissue respirometry on day 6 | day 6
  Oxidative Phosphorylation will be measured in muscle tissue using high resolution respirometry (Oroboros O2K) on day 6, after the 6 day methylpredinsolone treatment.
Expression level of NFKB Inducing Kinase (NIK) in tissue measured by real time PCR on day 0 | day 0
  NIK expression will be measured in muscle tissue using real time PCR on day 0.
Expression level of NFKB Inducing Kinase (NIK) in tissue measured by real time PCR on day 6 | day 6
  NIK expression will be measured in muscle tissue using real time PCR on day 6, after the 6 day methylprednisolone treatment.

SECONDARY OUTCOMES:
Lean Body Mass as measured by Dual Energy X-Ray Absorptiometry on day 0 | day 0
  Lean body mass will be measured using a Hologic DEXA on day 0.
Lean Body Mass as measured by Dual Energy X-Ray Absorptiometry on day 6 | day 6
  Lean body mass will be measured using a Hologic DEXA on day 6, after the 6 day methylprednisolone treatment.
Fat Mass as measured by Dual Energy X-Ray Absorptiometry on day 0 | day 0
  Fat mass will be measured using a Hologic DEXA on day 0.
Fat Mass as measured by Dual Energy X-Ray Absorptiometry on day 6 | day 6
  Fat mass will be measured using a Hologic DEXA on day 6, after the 6 day methylprednisolone treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Sheffield-Moore, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No